CLINICAL TRIAL: NCT05135728
Title: Development and Pilot Testing of a Novel Preschool Executive Function Curriculum Development of an Executive Function Intervention for Adolescents With Autism Spectrum Disorders
Brief Title: Development and Pilot Testing of a Novel Preschool Executive Function Curriculum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: AppleTree Institute (Unknown); The Maddux School (Unknown)
Responsible Party: Principal Investigator, Allison Ratto, Psychologist, Center for Autism Spectrum Disorders, Children's National Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00014103
Record Dates: First submitted 2021-10-06; First posted 2021-11-26 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Executive Dysfunction
Keywords: young children; intervention; preschool

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unstuck and On Target-Preschool (Experimental): UOT-P is based on the foundational principles of UOT for improving EF as well as evidence-based teaching methods (e.g., positive behavior supports, visual aids). Through this program, children, teachers and parents develop a shared self-regulatory vocabulary that enables children to improve EF at home and school through adult modeling and gradual scaffolding. The self-regulatory vocabulary (e.g., Flexible, Make a New Plan, Unstuck) becomes a "contagious" common language. We hypothesize this is the mechanism of change by which children will show improved EF skills, leading to increased academic readiness, improved social competence and reduced externalizing behaviors.
  Interventions: Behavioral: Unstuck and On Target: Preschool
- Waitlist Control (Active Comparator): Children at clinic sites beginning in Year 4 will be placed in Arm 2, in which a waitlist control model will be used. Assessment of participants on outcome measures will occur at pre-intervention, followed by a 16-week waitlist period, again at baseline, followed by a 16-week intervention, and then finally at endpoint. All participants in Arm 2 will receive UOT-P as their intervention (see Experimental Arm).
  Interventions: Behavioral: Unstuck and On Target: Preschool

INTERVENTIONS:
Behavioral: Unstuck and On Target: Preschool — Unstuck & On Target: Preschool (UOT:P) is a group-based curriculum for preschool and kindergarten students that targets executive function skills using CBT techniques. The UOT-P curriculum consists of 16 child small-group or classroom-wide lessons. Each lesson follows a clear structure in which the theme for the session is introduced in a storybook, supported with manipulatives and visuals. Children implement the skills introduced in the storybook through joing play activities that require them to flexibly adjusting their plans to work together. Children learn key vocabulary and active coping and problem-solving skills, with adult modeling and scaffolding, that enable them to build early executive functioning skills for self-regulation and classroom participation.

SUMMARY:
Executive function (EF) skills are a set of essential cognitive abilities that enable individuals to demonstrate their knowledge and talents, effectively complete tasks and navigate social interactions through flexible regulation of their thinking, behavior and emotions. EF is strongly linked to academic readiness and long-term educational outcomes. Children's EF is impacted by poverty-related experiences and is also impaired in the increasing number of children with developmental and emotional disabilities. Interventions targeting EF skills hold particular promise for improving children's educational trajectories by leveraging brain plasticity in the preschool period. We will directly target EF skills in preschoolers with poor EF. This project will address a key source of the achievement gap by meeting the needs of children at the highest risk, those who: 1) show early signs of EF impairment; 2) live in low-income communities and 3) are at risk for developmental and emotional disabilities (DD/ED). The intervention is a downward extension of Unstuck and On Target for elementary school (UOT; Cannon, Kenworthy, Alexander, Werner, & Anthony, 2018), an EF intervention shown to be effective at increasing children's learning behaviors, as delivered by school staff. The research team will partner with key stakeholders to revise and iteratively refine UOT-P through a development trial, utilizing participant, teacher and parent feedback. The results of this trial will be leveraged to enable the team to apply for future federal funding for a randomized comparative effectiveness trial (NIH, Institute of Educational Sciences, Patient-Centered Outcomes Research Institute).

ELIGIBILITY:
Inclusion Criteria:

Enrolled as a student at a participating school site OR as a patient at a participating clinic site

* Chronological age between 3-6 years at enrollment
* English as a primary language
* Roughly age-appropriate core language skills as determined by referring school staff or provider
* Identified by school staff or provider as having problems with flexibility

Exclusion Criteria:

No longer enrolled at participating school or clinic site

• Insufficient English fluency or language skills to complete intervention

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of Intervention | Through study completion, average of 20 weeks
  Interventionist ratings of feasibility will serve as the primary outcome measure. Interventionists will rate overall intervention feasibility using the Feasibility of Intervention Measure (FIM) at outcome. Scores range 4-20, where higher scores indicate higher feasibility.
Feasibility - Child Attendance | Through study completion, average of 20 weeks
  Child attendance at groups will also be tracked.
Acceptability of Intervention | Through study completion, average of 20 weeks
  Acceptability will be measured via interventionist ratings on the Acceptability of Intervention Measure (AIM). Scores range from 4-20, where higher scores indicate higher acceptability.
Intervention Appropriateness | Through study completion, average of 20 weeks
  Acceptability will be measured via interventionist ratings on the the Intervention Appropriateness Measure (IAM) at outcome.

SECONDARY OUTCOMES:
Fidelity Observations | twice throughout intervention period, average of 6 weeks between observations
  The Unstuck Treatment Implementation Measure will be used to assess interventionist fidelity. Standardized observations will be conducted, with ratings of fidelity on a Likert scale across several dimensions.
Interventionist Knowledge | baseline, end of intervention - an average of 20 weeks between baseline and end of intervention
  Interventionist knowledge of executive functioning and intervention strategies will be assessed using a five-item multiple-choice survey.

OTHER OUTCOMES:
Child Behavior Rating Scale (CBRS) | baseline, end of intervention - an average of 20 weeks between baseline and end of intervention
  This is a development trial, and thus primary outcomes assess feasibility and acceptability. However, preliminary investigation of child-level outcomes will also be undertaken. Classroom teachers will respond complete the CBRS, which uses a Likert scale to rate children's classroom behaviors for engagement with academic tasks, adults, and peers.
Head-Toes-Knees-Shoulders Revised (HTKS-R) | baseline, end of intervention - an average of 20 weeks between baseline and end of intervention
  This is a development trial, and thus primary outcomes assess feasibility and acceptability. However, preliminary investigation of child-level outcomes will also be undertaken. Trained assessors will administer the HTKS-R to child participants, which assesses self-regulation and emerging executive functioning. The HTKS-R is a short (5-8 minutes) behavioral task that assess children's working memory and impulse control through a short game in which children are introduced to paired body parts and instructed to touch the opposite body part of the one named.
Differential Ability Scales-II (DAS-II): Pattern Construction | baseline, end of intervention - an average of 20 weeks between baseline and end of intervention
  This is a development trial, and thus primary outcomes assess feasibility and acceptability. However, preliminary investigation of child-level outcomes will also be undertaken. The Pattern Construction subtest of the DAS-II will be administered to child participants. It requires children to replicate a visual design with blocks under timed conditions. Performance on this task is correlated with executive functioning abilities.
Classroom Observations | baseline, end of intervention - an average of 20 weeks between baseline and end of intervention
  This is a development trial, and thus primary outcomes assess feasibility and acceptability. However, preliminary investigation of child-level outcomes will also be undertaken. Trained evaluators will observe child participants' behavior over the course of 10-15 minutes in the classroom. Behaviors directly targeted in the intervention will be coded using a yes/no rating to indicate the presence or absence of a problem behavior during the observation.
Behavior Rating Inventory of Executive Functioning-Preschool (BRIEF-P): Selected subscales | baseline, end of intervention - an average of 20 weeks between baseline and end of intervention
  This is a development trial, and thus primary outcomes assess feasibility and acceptability. However, preliminary investigation of child-level outcomes will also be undertaken. Parent report of child participant behavior on the Shift and Emotional Control subscales of the BRIEF-P (an age-normed parent report measure of daily executive functioning problems in preschoolers) will be used to assess change in daily executive functioning skills.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Kenworthy, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No